CLINICAL TRIAL: NCT05425589
Title: Adjustable Strabismus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/2
Record Dates: First submitted 2022-03-29; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Intervention Model Description: Prospective, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjustable strabismus surgery (Other): Our objective was to assess the long-term success of adjustable suture strabismus surgery in terms of postoperative alignment and complications.
  Interventions: Procedure: Adjustable strabismus surgery

INTERVENTIONS:
Procedure: Adjustable strabismus surgery — Our objective was to assess the long-term success of adjustable suture strabismus surgery in terms of postoperative alignment and complications.

SUMMARY:
Strabismus, whether congenital or acquired, is a common visual and cosmetic problem, especially for the young. Adjustable suture strabismus surgery is not in vogue in our country. This technique gives the surgeon a second attempt to provide a better outcome for the patients.

ELIGIBILITY:
Horizontal, vertical and complex strabismus cases (sensory, paralytic, nystagmus, monocular elevation deficit and dissociated vertical/horizontal deviation) were included, along with patients with a previous history of strabismus surgery.

Myasthenia gravis was excluded along with noncooperative children; less than 7 years of age. Those who did not return for a one year follow up also had to be excluded.

Ages: 5 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative alignment | 1 year
  The post-operative alignment at 1 year will be measured and compared with the pre-operative alignment (deviation) to assess success rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan